CLINICAL TRIAL: NCT01831960
Title: An Open Label Evaluation of the Adrenal Suppression Potential and Pharmacokinetic Properties of Cortexolone 17α-Propionate (CB-03-01) Cream Applied Every Twelve Hours for Two Weeks in Subjects With Acne Vulgaris
Brief Title: An Evaluation of the Adrenal Suppression Potential and Pharmacokinetic Properties of CB-03-01 Cream in Subjects With Acne Vulgaris
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Intrepid Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 171-7151-202
Record Dates: First submitted 2013-04-11; First posted 2013-04-15 (Estimated); Results first posted 2020-11-17 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-11

CONDITIONS: Acne Vulgaris
Keywords: Cassiopea; clascoterone; cortexolone 17α-propionate; anti-androgen; CB-01-03
MeSH Terms: conditions — Acne Vulgaris | interventions — Clascoterone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cortexolone 17α-Propionate (Experimental): Topical cream, 1.0% concentration, applied every twelve hours
  Interventions: Drug: cortexolone 17α-propionate

INTERVENTIONS:
Drug: cortexolone 17α-propionate
  Other Names: CB-03-01; clascoterone (USAN, INN)

SUMMARY:
This study is designed to determine the hypothalamic-pituitary-adrenal (HPA) axis suppression potential and pharmacokinetic (PK) properties of CB-03-01 Cream, 1%, applied every twelve hours for two weeks, in subjects with acne vulgaris ages 12 years or older.

ELIGIBILITY:
Inclusion Criteria:

* Subject has moderate to severe facial acne vulgaris as determined by the Investigator's Global Assessment (IGA) and obvious acne on the chest and/or back at study start.
* Subject has facial acne vulgaris (including the nose) with a minimum number of inflammatory lesions (papules, pustules, and nodules/cysts) and a minimum number of non-inflammatory lesions (open and closed comedones) at study start.
* Females must be post-menopausal, surgically sterile or using highly effective birth control methods with a negative urine pregnancy test (UPT) at study start.
* Subject must be in general good health in the opinion of the investigator, with normal renal function, based on screening physical examination, medical history, and clinical laboratory values.

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject is 12-20 years of age and has a Body Mass Index (BMI) for age percentile > 85%.
* Subject is > 20 years of age and has a BMI > 32.0 kg/m2.
* Subject has used tobacco, smoking cessation products, or products containing nicotine within three months prior to study start.
* Except for the use of contraceptives, subject has used any prescription drug or herbal product within 14 days prior to dosing, any non-prescription drug or vitamin or mineral supplements within 7 days prior to study start; any known enzyme-inducer, enzyme-inhibitor, or reported chronic exposure to enzyme-inducers such as paint solvents or pesticides within 30 days of study start.
* Subject has used topical anti-acne medications containing retinoids such as tazarotene, adapalene or tretinoin, within four weeks of study start.
* Subject has used the following systemic anti-acne medications: antibiotics within two weeks of study start, spironolactone within four weeks of study start, or retinoid therapy within three months of study start.
* Subject has any skin or medical condition, including facial hair that could interfere with the evaluation of the test article or requires the use of interfering topical or systemic therapy.
* Subject has the need or plans to be exposed to artificial tanning devices or excessive sunlight during the study.
* Subject has used light treatments, microdermabrasion or chemical peels to the face, chest and back within eight weeks of study start.
* Subject cannot avoid any type of strenuous exercise (swimming, running, team sports, etc.,) or the use of hot tubs/saunas from study start to the end of the study.
* Subject has received an investigational drug or been treated with an investigational device within 30 days prior to study start.
* Subject is currently enrolled in an investigational drug or device study.
* Subject has used topical corticosteroids (including inhaled and intranasal corticosteroids) within two weeks of study start.
* Subject has used systemic corticosteroids (including intramuscular and intralesional injections) within four weeks of study start.
* Subject has an irregular sleep schedule or works night shifts.
* Subject has experienced significant blood loss within 60 days or has donated plasma within 72 hours prior to study start.
* Subject tests positive at Screening for human immunodeficiency virus (HIV) or is known to be seropositive for HIV.
* Subject tests positive at Screening for hepatitis B surface antigen, hepatitis C antibody or has a history of a positive result.
* Subject had major surgery within 30 days prior to study start or plans to have surgery during the study.
* Subject has participated in a previous CB-03-01 study.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-04; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: R&D Cassiopea, Study Director — Cassiopea S.p.A.
Locations (3):
- United States (3):
  - Northwest Clinical Trials, Inc., Boise, Idaho
  - Shideler Clinical Research Center, Carmel, Indiana
  - Michigan Center for Research Corp., Clinton Township, Michigan

RESULTS

PARTICIPANT FLOW:
Groups:
- Cortexolone 17α-Propionate (Cohort 1): Cohort 1 enrolled adult subjects. Topical cream, 1.0% concentration, applied every twelve hours.
- Cortexolone 17α-Propionate (Cohort 2): Cohort 2 enrolled adolescent subjects 12 to less than 18 years of age. Topical cream, 1.0% concentration, applied every twelve hours.
Period: Overall Study
Arm/Group | Cortexolone 17α-Propionate (Cohort 1) | Cortexolone 17α-Propionate (Cohort 2)
Started | 20 | 22
Completed | 20 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Forty-two (42) subjects were enrolled into the study across two cohorts dependent upon age:
  Cohort 1: 20 adult subjects Cohort 2: 22 adolescent (12 to less than 18 years of age) subjects
Groups:
- Cortexolone 17α-Propionate (Cohort 1): Topical cream, 1.0% concentration, applied every twelve hours.
- Total: Total of all reporting groups
Arm/Group | Cortexolone 17α-Propionate (Cohort 1) | Cortexolone 17α-Propionate (Cohort 2) | Total
Number analyzed (Participants) | 20 | 22 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Forty-two (42) subjects were enrolled into the study across two cohorts dependent upon age:
  Cohort 1: 20 adult subjects Cohort 2: 22 adolescent (12 to less than 18 years of age) subjects
  years | 24.4 (5.84) | 15.6 (1.33) | 19.8 (6.02)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: See note above.
  Participants
    Female | 15 | 12 | 27
    Male | 5 | 10 | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: See note above.
  Participants
    Hispanic or Latino | 0 | 1 | 1
    Not Hispanic or Latino | 20 | 21 | 41
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: See note above.
  Participants
    American Indian or Alaska Native | 0 | 0 | 0
    Asian | 1 | 0 | 1
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 1 | 0 | 1
    White | 17 | 21 | 38
    More than one race | 1 | 1 | 2
    Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in HPA Axis Response to Cosyntropin
Description: Measurement of serum cortisol concentrations after stimulation of the adrenal cortex with cosyntropin injection (Cosyntropin Stimulation Test - CST). Prior to CST, a pre-CST blood sample is taken between 7AM to 9AM. Thirty minutes after CST, a post-CST blood sample is collected. HPA axis suppression is defined as a post-stimulation serum cortisol level ≤ 18 μg/dL at Day 14.
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: mcg/dL
Groups:
- Cortexolone 17α-Propionate (Cohort 1): Cohort 1 enrolled adults subjects. Topical cream, 1.0% concentration, applied every twelve hours.
Arm/Group | Cortexolone 17α-Propionate (Cohort 1) | Cortexolone 17α-Propionate (Cohort 2)
Number analyzed (Participants) | 20 | 22
mcg/dL
  Baseline (pre-CST) | 17.0 (5.98) | 16.8 (4.71)
  Baseline (post-CST) | 27.7 (3.43) | 24.6 (3.12)
  Day 14 (pre-CST) | 18.1 (7.02) | 15.4 (3.98)
  Day 14 (post-CST) | 26.7 (5.56) | 22.8 (2.99)

2. Primary Outcome: PK Profiles (Cmax) of Cortexolone 17α-propionate
Description: Max concentration (Cmax) of cortexolone 17α-propionate in plasma following the first application (i.e., Day 1, 0-12 hours) and last application (i.e., Day 14, 0-12 hours).
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cortexolone 17α-Propionate (Cohort 1) | Cortexolone 17α-Propionate (Cohort 2)
Number analyzed (Participants) | 20 | 22
ng/mL
  Cmax - Day 1 (ng/mL) | 3.23 (2.01) | 3.58 (4.30)
  Cmax - Day 14 (ng/mL) | 4.46 (3.00) | 4.61 (4.74)

3. Primary Outcome: PK Profiles (AUC) of Cortexolone 17α-propionate
Description: Area under the plasma concentration curve (0-12 hours) of cortexolone 17α-propionate at baseline (i.e., Day 1, after first application [0-12 hours]) and at Day 14 (i.e., Day 14, after last application [0-12 hours]).
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Cortexolone 17α-Propionate (Cohort 1) | Cortexolone 17α-Propionate (Cohort 2)
Number analyzed (Participants) | 20 | 22
hr*ng/mL
  AUCτ - Day 1 | 22.02 (13.67) | 22.55 (22.57)
  AUCτ - Day 14 | 37.14 (22.92) | 30.97 (24.65)

4. Primary Outcome: PK Profiles (Cavg) of Cortexolone 17α-propionate
Description: Average concentration of cortexolone 17α-propionate in plasma calculated as the ratio of the AUC(0-12 hours) and the dosing interval (i.e., 12 hours) at baseline (i.e., Day 1, after first application) and at Day 14 (after last application).
Time Frame: Baseline and Day 14
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Cortexolone 17α-Propionate (Cohort 1) | Cortexolone 17α-Propionate (Cohort 2)
Number analyzed (Participants) | 20 | 22
ng/mL
  Cavg - Day 1 | 1.84 (1.14) | 1.88 (1.88)
  Cavg - Day 14 | 3.10 (1.91) | 2.58 (2.05)

ADVERSE EVENTS:
Time Frame: 14 Days
Description: Any treatment emergent AEs ongoing at the end of the treatment period (Day 14) were followed until they resolve, the condition stabilizes, the events are otherwise explained, or the subject is lost to follow-up. In addition, all SAEs were followed until resolution as previously stated for study product-related AEs.
Arm/Group | Cortexolone 17α-Propionate (Cohort 1) | Cortexolone 17α-Propionate (Cohort 2)
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/22
Other Adverse Events (participants affected / at risk) | 5/20 | 3/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cortexolone 17α-Propionate (Cohort 1) (N=20) | Cortexolone 17α-Propionate (Cohort 2) (N=22)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Application site folliculitis (General disorders) | 1 (1) | 0 (0)
Ear infection (Infections and infestations) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
ACTH stimulation test abnormal (Investigations) | 1 (1) | 2 (2) — Adrenocorticotropic Hormone (ACTH) stimulation testing is conducted by the Cosyntropin Stimulation Test.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Sponsor has first right to publish pooled study data. In the event that such manuscript has not been submitted for publication within 18 months from study completion/termination at all participating sites, the PI shall have the right to single center publications provided they submit any data for presentation, oral or written, to the Sponsor for review 60 days prior to public disclosure. The PI may not disclose previously undisclosed confidential information other than study results.